CLINICAL TRIAL: NCT04640831
Title: A Phase 1 Dose-ranging Study of GH001 in Healthy Volunteers
Brief Title: Safety of GH001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GH001-HV-101; 2018-003632-68 (EudraCT Number)
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; 5-MeO-DMT; 5-methoxy-dimethyltryptamine
MeSH Terms: interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Intervention Model Description: Part A: Dose ranging in four dose groups Part B: One group with individualized dosing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GH001 dose A (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- GH001 dose B (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- GH001 dose C (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- GH001 dose D (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- GH001 Individualized Dosing (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine

INTERVENTIONS:
Drug: 5 Methoxy N,N Dimethyltryptamine — GH001 administered via inhalation
  Other Names: GH001; 5-MeO-DMT

SUMMARY:
The aim of the study is to investigate the safety of GH001 (containing 5-methoxy-dimethyltryptamine; 5-MeO-DMT), and its dose-related psychoactive effects in healthy volunteers.

The study will evaluate single, ascending doses of GH001 in Part A and an individualized dosing regimen of GH001 in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) in the range of 18.5 and 27.0 kg/m2 (inclusive);
* Subject is in good general health in the opinion of the medical supervisor;
* Subject is in good mental health in the opinion of the (clinical) psychologist as determined by the intake interview;

Exclusion Criteria:

* Has known allergies or hypersensitivity or any other contraindication to 5-MeO-DMT;
* Has received any investigational medication within the last 1 month.
* Has a medically significant condition, which renders the subject unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of GH001 | up to 7 days
  The safety and tolerability of GH001 is judged by the Study Safety Group based on a combined analysis of reported adverse events, clinical observation, and safety laboratory analyses.
The dose-related psychoactive effects of GH001 as evaluated by a Visual Analogue Scale | Retrospectively assessed at 3 hours
  Visual Analogue Scale scored from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: GH Research Clinical Team, Study Director — GH Research Ireland Limited
Locations (1):
- Clinical Trial Site, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reckweg J, Mason NL, van Leeuwen C, Toennes SW, Terwey TH, Ramaekers JG. A Phase 1, Dose-Ranging Study to Assess Safety and Psychoactive Effects of a Vaporized 5-Methoxy-N, N-Dimethyltryptamine Formulation (GH001) in Healthy Volunteers. Front Pharmacol. 2021 Nov 25;12:760671. doi: 10.3389/fphar.2021.760671. eCollection 2021. PMID 34912222